CLINICAL TRIAL: NCT05125770
Title: Study on the Safety of New Coronavirus Vaccination for Couples During the Peri-pregnancy Period on the Fetus
Brief Title: Study on the Fetal Safety of New Coronavirus Vaccination for Couples During the Peri-pregnancy Period
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Ditan Hospital (Other)
Responsible Party: Principal Investigator, Wei Yi, Director, Head of Obstetrics and Gynecology, Beijing Ditan Hospital
Other Study IDs: KY2021-12
Record Dates: First submitted 2021-11-08; First posted 2021-11-18 (Actual); Last update posted 2021-11-18 (Actual); Status verified 2021-11

CONDITIONS: Perinatal
Keywords: propofol tenofovir; HBV DNA; mother-to-child block; New crown vaccination; Perinatal period

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- new crown vaccination: Collect all the couples who gave birth in Ditan Hospital or one of the mothers and newborns who were injected with the new crown vaccine during the peri-pregnancy period as the observation group
  Interventions: Biological: New crown vaccine
- non new crown vaccination: Collect the pregnant women and newborns who were not vaccinated with the new crown vaccine during the peri-pregnancy of the couples who gave birth in our hospital during the same period as the control group

INTERVENTIONS:
Biological: New crown vaccine — New Coronavirus vaccine
  Groups: new crown vaccination

SUMMARY:
All the pregnant women and newborns of both or one of the couples who gave birth in Ditan hospital were collected as the observation group, and the pregnant women and newborns of both husband and wife who gave birth in our hospital without new crown vaccine during pregnancy were collected as the control group. The incidence of adverse events during pregnancy of the two groups and the incidence of intrauterine development and congenital malformations of the two groups were observed to observe the physical and intellectual development of children in the two groups at the age of 1 year, and to explore the safety of perinatal neocrown vaccination.

DETAILED DESCRIPTION:
This study is a prospective observational cohort study. All the pregnant women and newborns of both or one of the couples who gave birth in Ditan hospital were collected as the observation group, and the pregnant women and newborns of both husband and wife who gave birth in our hospital without new crown vaccine during pregnancy were collected as the control group. The incidence of adverse events during pregnancy of the two groups and the incidence of intrauterine development and congenital malformations of the two groups were observed to observe the physical and intellectual development of children in the two groups at the age of 1 year, and to explore the safety of perinatal neocrown vaccination.

ELIGIBILITY:
Inclusion Criteria:

* The pregnant women and newborns who were injected with the new crown vaccine during the perinatal period of both husband and wife or one of them were the observation group, and the pregnant women and newborns who were not vaccinated with the new crown vaccine during the perinatal period of both husband and wife were the control group. They were fully informed of the risk, voluntarily joined the study and signed the informed consent.

Exclusion Criteria:

* Both husband and wife or family have previously delivered congenital abnormal fetus;
* Neither husband nor wife was willing to participate in this study.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The pregnant women and newborns who were injected with the new crown vaccine during the perinatal period of both husband and wife or one of them were the observation group, and the pregnant women and newborns who were not vaccinated with the new crown vaccine during the perinatal period of both husband and wife were the control group. They were fully informed of the risk, voluntarily joined the study and signed the informed consent.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-11-08 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Neonatal congenital malformation rate | at birth
  Observe whether the newborn has malformation
Intellectual development of 1-year-old children | at one year old
  The intellectual development of newborns was observed

SECONDARY OUTCOMES:
Incidence of maternal adverse events during pregnancy | during pregnancy
  Observe the incidence of maternal adverse events during pregnancy
Physical development of children at birth and 1 year old | at birth, at 1 year old
  Observe the physical development of children at birth and 1 year old
The incidence of adverse events among children aged 1 year | among 1 year old
  Observe the incidence of adverse events among children aged 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Ditan Hospital, Capital Medical University, Beijing, Beijing Municipality, China